CLINICAL TRIAL: NCT00579163
Title: Ascertainment of Peripheral Blood or Saliva Samples for Genetic Epidemiology Studies of Familial Cancers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 93-102
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Uterine Cervical Neoplasms; Leukemia; Lymphoma, Non-Hodgkin
Keywords: Blood; Salvia; Tissue
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Prostatic Neoplasms; Uterine Cervical Neoplasms; Leukemia; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Saliva, Tumor Tissue, Normal Tissue

SUMMARY:
The purpose of this study is to better understand the genetic causes of cancer and the inherited tendency to develop cancer. To accomplish this, blood specimens and/or saliva samples and/or tumor and normal tissue blocks from patients and families of patients with cancer will be collected. Blood specimens will be frozen and stored for analysis at a later date. Tumor tissue and normal tissue will be stored for analysis at a later date. In order to perform this study, patients and members of their families will be asked to provide blood samples and/or saliva samples. Individuals will be asked to provide a history of cancer in their relatives at the time the blood sample is given. No relatives will be contacted before they have been asked by a family member if they wish to participate in this study. If they do wish to participate, the relatives should indicate this by returning the "Family Member Consent for Contact Form" After we receive this form, arrangements may be made for the family member to send in a blood and/or saliva sample or to come in person to provide the sample to us.

Except for family history, no medical information provided by one member of a family will be discussed with other family members. At the end of this form, we will also ask for your permission to be contacted in the future to discuss information about your health, additional research with your samples and/or certain research findings possibly related to your sample.

DETAILED DESCRIPTION:
Patients can provide either a blood or saliva sample for the protocol. For blood samples, two tubes of blood (approximately 20 cc) will be drawn from the patient, utilizing a sterile technique. The tubes will be rocked so as to mix the blood with the additive (EDTA) in the tubes. For saliva samples, approximately 2-4 ml of saliva will be collected in specialized Oragene DNA Self-Collection Kit tubes. The sample(s) may also be used to detect new genes or changes in genes that may tell us who is at risk for certain types of cancer and/or other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for referral to the Cancer Family Clinic of the Department of Medicine at Memorial Sloan-Kettering Cancer Center are eligible for participation in this study. Such patients should have a history of cancers of the breast, ovary, colon, prostate, uterus, non-Hodgkin's lymphoma, leukemia, soft tissue sarcoma, endocrine neoplasms, or other malignancies presenting in first degree relatives or in successive generations as part of a suspected cancer family syndrome.
* Family members of probands including parents, sisters, brothers, half-brothers and sisters, sons, daughters, grandparents, as well as aunts and uncles are also eligible.
* This study involves research which presents no greater than minimal risk to children. The assent of any minor should be obtained before the patient is entered into this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 992 (Actual)
Dates: Start 1994-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To establish a bank of DNA and frozen lymphoblastoid cell lines for the purpose of facilitating genetic epidemiology investigations of familial cancers. | 1 year

SECONDARY OUTCOMES:
A related goal is to provide patients with cancer and their living relatives the opportunity to preserve DNA samples so that they may be used for future genetic counseling regarding inherited cancer risk. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT00579163/ICF_000.pdf